CLINICAL TRIAL: NCT04698265
Title: Comparison of the Efficacy of Intra-articular Injection of Human Amniotic Suspension Allograft and Platelet-rich Plasma in the Treatment of Knee Osteoarthritis: A Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Efficacy of Intra-articular Injection of Human Amniotic Suspension Allograft and Platelet-rich Plasma in the Treatment of Knee Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yin Ming, Huang, Chief resident of Orthopedic., Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KSVGH20-CT9-11, ASA RCT 1.0
Record Dates: First submitted 2020-12-20; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Human amniotic suspension allograft (ASA), 40 mg (Experimental): Human amniotic suspension allograft (ASA) contains particulated human amniotic membrane and cells derived from the amniotic fluid. The allograft is freeze-dried, terminally sterilized with low dose gamma irradiation. Arm 1 uses 40 mg ASA stored in a sterile vial (Amniogen, HTC Regenerative Ltd. New Taipei, Taiwan).
  Interventions: Biological: Human amniotic suspension allograft (ASA)
- Human amniotic suspension allograft (ASA), 20 mg (Experimental): Human amniotic suspension allograft (ASA) contains particulated human amniotic membrane and cells derived from the amniotic fluid. The allograft is freeze-dried, terminally sterilized with low dose gamma irradiation. Arm 2 uses 20 mg ASA stored in a sterile vial (Amniogen, HTC Regenerative Ltd. New Taipei, Taiwan).
  Interventions: Biological: Human amniotic suspension allograft (ASA)
- CellularMatrix (a combination of platelet-rich plasma and hyaluronic acid) (Experimental): CellularMatrix (RegenLab SA, Switzerland) is composed of sterile and non-pyrogenic tubes allowing the mix of Platelet Rich Plasma (PRP) with Hyaluronic Acid (HA) in the same proportion (2mL of PRP for 2mL of HA).
  Interventions: Biological: Human amniotic suspension allograft (ASA)
- Normal saline (Placebo Comparator): 4ml of normal saline
  Interventions: Biological: Human amniotic suspension allograft (ASA)

INTERVENTIONS:
Biological: Human amniotic suspension allograft (ASA) — Human amniotic suspension allograft (ASA) intra-articular injection.

SUMMARY:
A double-blind, randomized controlled trial designed to evaluate the symptomatic modulating efficacy of amniotic suspension allograft (ASA) in comparison to platelet-rich plasma (PRP), hyaluronic acid (HA) and normal saline (NS) in the injection treatment of knee osteoarthritis. The hypothesis is that ASA would provide the greatest functional improvement.

DETAILED DESCRIPTION:
At least 150 subjects with osteoarthritic knee will be recruited and computer randomized 1:1:1:1 to single injection of ASA (40mg), ASA (20mg), PRP + HA, and NS groups. Both subjects and evaluaters were blinded to allocations. Functional and radiologic outcomes were measured at baseline, and 1 week, 1, 3, 6, 12 months postinjection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years
* Ability to provide informed consent
* Unilateral or bilateral knee VAS pain score ≥ 4 of 10 (worst possible pain) for more than 4 months
* Diagnosis of OA Kellgren-Lawrence I-III by radiography (triple-film of bilateral lower limb, standard knee anterior-posterior view in full extension, lateral view in 30-degrees flexion, and 45°Merchant views)
* No prior PRP injection of knee
* No prior surgical procedure of the participating knee
* BMI<40 kg/m2

Exclusion Criteria:

* Lawrence stage IV
* Major axial deviation (varus> 5°, valgus > 5°)
* Any concomitant symptomatic knee disorder (i.e. ligamentous/ meniscal injury)
* Systemic inflammatory arthropathy
* Hematologic diseases
* Severe cardiovascular disease
* Neurological disorders
* Active infection
* Immuno-compromised
* Therapy with anticoagulants or antiaggregants
* Use of NSAIDs and/or chondroprotective supplements, such as glucosamines and chondroitin sulfates, within 7 days prior to trial
* Recent intra-articular injection of corticosteroids (within 30 days)
* Prior treatment with HA in past 6 monthsHb< 11 g/dL
* Platelet count < 150,000/mm3

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) between baseline, 1 week, and 1 ,3 ,6 ,12 months. | Baseline, 1 week, 1,3,6,12 months
  WOMAC is a self-administered questionnaire consisting of 24 items divided into 3 subscales:(1) Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright(2) Stiffness (2 items): after first waking and later in the day(3) Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic dutiesThe test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).

SECONDARY OUTCOMES:
Change of the International Knee Documentation Committee (IKDC Questionnaire) between baseline, 1 week, and 1 ,3 ,6 ,12 months. | Baseline, 1 week, 1,3,6,12 months
  The International Knee Documentation Committee Questionnaire is a knee-specific patient-reported outcome measure.The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Meanwhile, the sports activity subscale focuses on functions like going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks patients one simple question: how is their knee at present versus how was their knee prior to injury? Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100, This final number is interpreted as a measure of function with higher scores representing higher levels of function.

IPD SHARING:
Plan to Share IPD: No
We do not have the plan to make individual participant data (IPD) available to other researchers.